CLINICAL TRIAL: NCT05840965
Title: Differences in Foot Biomechanics and the Effect of Foot Core Exercises or Foot Orthotics in Symptomatic Flexible Flatfoot
Brief Title: The Effect of Foot Core Exercises or Foot Orthotics in Symptomatic Flexible Flatfoot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Nicolas Haelewijn, Physiotherapist, Master of Science, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B3222022001031; S67036 (Other: KU Leuven, Belgium)
Record Dates: First submitted 2023-03-03; First posted 2023-05-03 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Flatfoot, Flexible
Keywords: Multi segment foot kinetics; Multi segment foot kinematics; Intrinsic foot muscles; Ultrasound
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Intervention Model Description: Prospective monocentric randomised controlled trial with an asymptomatic control group.
Who Masked: Outcomes Assessor
Masking Description: The data will be coded (pseudonymization). The subject's name or other identifiers will be stored separately from their research data and replaced with a unique code to create a new identity for the subject.
  The outcomes assessor will be blind for participants' injury status for the following :
  * while conducting kinematic and kinetic data processing,
  * while performing muscle size measurements on the ultrasound images,
  * while performing statistical analysis (for all outcomes)
  There will be no blinding while scoring the following outcomes (because these scores are immediately determined in the presence of the participant) :
  * Foot muscle strength
  * Foot posture index
  * Navicular drop
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Asymptomatic flexible flatfoot (No Intervention): This group undergoes no intervention.
- Symptomatic flexible flatfoot: foot core strengthening (Experimental): The investigators put together a specific training program emphasizing the neuromuscular recruitment of the plantar intrinsic foot muscles. This will be colloquially referred to as the "Foot Core Strengthening Program". The most recognized exercise of our program is the short foot exercise. However, as recently other exercises were validated by Gooding et al., we also included following exercises: toe spread out, first-toe extension and second- to fifth-toes extension. Simultaneously, neuromuscular electrical stimulation (NMES) will be provided, as 77% of healthy active people struggle performing contractions of the foot muscles.
  Interventions: Other: Foot muscle strengthening
- Symptomatic flexible flatfoot: foot orthotics (Active Comparator): Custom-made foot orthotics are the current standard of care (SOC) therapy within this population. Patients choose their own health care provider to customize these orthotics. The sole is made of EVA material whose color and hardness is determined by the podiatrist or bandage maker. Digital scans or plaster of Paris cast will be taken of the participant's non-weightbearing foot (placed in a neutral or corrected position) by a certified pedorthist following the prescription of the orthopaedic surgeon.
  The geometry of the foot orthotic will encompass a total contact principle with respect to the medial arch. The orthotics will be manufactured using ethyl vinyl acetate (EVA) with a shore ranging between 45 and 60
  Interventions: Other: Foot orthotics

INTERVENTIONS:
Other: Foot muscle strengthening — A specific training program emphasizing the neuromuscular recruitment of the plantar intrinsic foot muscles. This will be colloquially referred to as the "Foot Core Strengthening Program". The exercises are: short foot exercise, toe spread out, first toe extension, second to fifth toe extension. Simultaneously, neuromuscular electrical stimulation (NMES) will be provided, as 77% of healthy active people struggle performing contractions of the foot muscles.
  Arms: Symptomatic flexible flatfoot: foot core strengthening
Other: Foot orthotics — Custom-made foot orthotics
  Arms: Symptomatic flexible flatfoot: foot orthotics

SUMMARY:
The overall goal of this study is to evaluate the effect of a foot strengthening program (focused on the intrinsic foot muscles) on ankle and foot joint kinematics and kinetics (rearfoot, midfoot, and forefoot) in patients with symptomatic flexible flat feet. The investigators will also evaluate the effect on intrinsic muscle morphology, foot strength, pain and other symptoms. The investigators will compare to the standard conservative therapy, which is foot orthotic therapy.

DETAILED DESCRIPTION:
A common condition is "symptomatic flexible flat foot". This clinical entity affects 1 in 5 adults and is characterized by misalignment of the foot joints, resulting in a flat medial longitudinal foot arch. As a result, the foot's load-bearing capacity is reduced, leading to overuse injuries such as back pain, patellofemoral pain, or medial tibial stress syndrome.

The literature shows that people with flexible flat feet have disturbed foot and ankle kinematics during locomotor tasks. However, the current literature lacks insight into the kinetics of the foot joints (i.e., forces that cause joint movement) during both relatively simple tasks such as walking and running and more challenging tasks such as landing from a step. The recent development of multisegmental kinetic foot models allows for detailed information to be obtained regarding (mal)adaptive joint loading patterns in this population and address shortcomings in the current literature.

In recent years, the small intrinsic foot muscles (IFM) have received more attention in the treatment of foot and ankle-related overuse injuries, such as plantar fasciitis, medial tibial stress syndrome, and Achilles tendinopathy. According to the "foot core" paradigm, the primary role of the intrinsic foot muscles is to support the medial foot arch. They contribute to the absorptive and generative capacity of the medial foot arch and work together with the plantar aponeurosis, ligaments, and extrinsic foot muscles. It is known that their strength and volume are reduced in people with flat feet.

A randomized controlled trial will be planned in which participants with symptomatic flexible flatfeet will be allocated to either receiving foot core strengthening exercises or custom made foot orthotics therapy. An asymptomatic group with flexible flatfeet will serve as a control group and will not undergo any intervention.

Primary objective 1: To evaluate changes in foot joint kinetics and kinematics and intrinsic foot muscle size following a foot core strengthening program in participants with symptomatic flexible flatfoot and whether this is different to the control therapy.

Secondary objective 1: To evaluate changes in foot posture, foot muscle strength, psychological scores, pain and symptoms following a foot core strengthening program and whether these changes are different in comparison to the control therapy.

Secondary objective 2: To evaluate changes in foot joint kinematics and kinetics and intrinsic foot muscle size between participants with asymptomatic and symptomatic flexible flatfoot.

ELIGIBILITY:
Inclusion Criteria:

For both asymptomatic and symptomatic flexible flatfoot:

* Adults between 18 and 65 years of age, able to run at a self- selected low speed.
* Physically active: min. 1h30 and max 6 h/week
* Foot Posture Index > 6 AND Navicular drop > 5 mm
* Informed consent (ICF) obtained

For asymptomatic flexible flatfoot:

cfr. supra

For symptomatic flexible flatfoot:

* Diagnosis made by a physician
* ICF obtained
* Symptomatic =
* Foot pain ( > 4 on Visual Analog Pain Scale score) OR
* Medial arch pain OR
* Metatarsalgia (general or diffuse hyperkeratosis accepted) OR
* Lateral impingement pain OR
* Sinus tarsi pain OR
* Tibialis posterior dysfunction stage I and II (without indication of rupture) and painful single heel raise test

Exclusion Criteria:

For both groups:

* < 18 years, > 65 years
* Any medical contraindication to physical exertion
* Systemic diseases
* Recent lower limb surgery (< 6 months)
* Lower limb osteosynthesis material
* Pregnancy
* Pacemaker
* Leg length discrepancy > 3 cm
* Body Mass Index (BMI) > 30kg/m²
* Constant ankle pain
* Ankle fractures
* Single hyperkeratotic lesion with nucleus under metatarsal head
* Recent participation in a physical rehabilitation program (< 3 months)
* Recent orthotics (< 3 months)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Change in lower limb joint angles (degrees) | 8-week intervention period
  Joint angles will be measured based on the position of passive markers placed on participants' anatomical landmarks all over the lower limbs. The position of those markers will be tracked by 10 infrared high-speed cameras that surround the walkway (sampled at 100 Hertz (Hz) - type T-10, 1 megapixel, captures 10-bit grayscale using 1120 * 896 pixels, Vicon Motion System Ltd, Oxford, Metrics, UK).
  The angular positions of the multiple joints that constitute the lower limb (hip, knee, ankle, chopart, lisfranc and metatarsophalangeal) will be assessed during walking, running, and single leg drop jump in the gait laboratory.
Change in lower limb joint angular velocities (degrees/second) | 8-week intervention period
  Joint angular velocities are also assessed based on reflexive markers placed on anatomical landmarks. This outcome evaluates the rate of change of a certain joint angle over time.
  Joint angular velocities will be assessed of the multiple joints that constitute the lower limb (hip, knee, ankle, chopart, lisfranc and metatarsophalangeal) during walking, running and a single leg drop jump in the gait laboratory.
Change in joint moments | 8-week intervention period
  Joint moments will be determined by coupling kinematic data (joint position and velocities) with plantar pressure data from a specially designed pressure plate (sampled at 200Hz, Footscan, dimension 0.5m x 0.4m, 4096 sensors, 2.8 sensors/cm², RsScan International, Olen, Belgium) embedded in the middle of the runway and placed on top of a force plate (sampled at 1000Hz, Advanced Mechanical Technology Inc., Watertown, MA, USA). Kinetic data will be assessed while walking, running and a single leg drop jump in the gait laboratory.
Change in foot muscle thickness | 8-week intervention period
  The thickness of five intrinsic foot muscles (abductor hallucis, flexor digitorum brevis, flexor hallucis, quadratus plantae and abductor digiti minimi) and three extrinsic foot muscles (peronei, tibialis anterior and flexor digitorum longus) will be measured on images obtained using ultrasonography.
  To obtain those images, the investigators will scan the muscles in a longitudinal view.
Change in foot muscle cross-sectional area | 8-week intervention period
  The area of five intrinsic foot muscles (abductor hallucis, flexor digitorum brevis, flexor hallucis, quadratus plantae and abductor digiti minimi) and two extrinsic foot muscles (peronei and flexor digitorum longus) will be measured on images obtained using ultrasonography.
  To obtain those images, the investigators will scan the muscles in a transversal view.

SECONDARY OUTCOMES:
Change in foot muscle strength | 8-week intervention period
  Foot muscle strength will be evaluated using a hand-held dynamometer, with participants hook lying. The investigators will both report the strength of the big toe and the strength of the other toes (as a whole).
Change in foot Posture Index | 8-week intervention period
  The Foot Posture Index 6-item is a validated six-item criterion reference tool for quantifying standing foot posture and is used in a variety of clinical and research settings 33. It is a quick and reliable tool to quantify the degree to which a foot is pronated, neutral or supinated. The patient stands in a relaxed stance position with double limb support while the assessor evaluates a total of 6 items via observations and palpations.
Change in navicular drop | 8-week intervention period
  The investigators will assess navicular drop as the difference in distance between the navicular tuberosity to the ground from sitting to double-limb stance.
Change in the OSPRO-YF questionnaire | 8-week intervention period
  The OSPRO-YF questionnaire will be used to assess individual psychological scores, including: depressive symptoms, anxiety, anger, fear-avoidance beliefs, kinesiophobia, catastrophizing, self-efficacy, and pain acceptance 32. This questionnaire is designed to evaluate multiple psychological scores without burdening a person with completing each full instrument.OSPRO-YF summarizes 11 psychological questionnaires, quartile scores are used instead of cutoff scores for consistency and assessment of a wide range of outpatient orthopedic patients.
Change in the FAOS questionnaire | 8-week intervention period
  The Foot and Ankle Outcome Score is a patient reported instrument useful for assessing changes in foot/ankle pathology over time with or without treatment. The score assesses pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and foot/ankle related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible foot/ankle symptoms and 100 indicating no foot/ankle symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Deschamps, PhD, Pod, Principal Investigator — Musculoskeletal Rehabilitation Research Group, Department of Rehabilitation Sciences, KU Leuven
Locations (1):
- KU Leuven, Bruges, West Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No